CLINICAL TRIAL: NCT01397539
Title: A Randomized, Blinded, Placebo-Controlled Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB037 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Single Ascending Dose Study of BIIB037 in Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 221AD101
Record Dates: First submitted 2011-06-30; First posted 2011-07-19 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIIB037 (Experimental): A single dose of BIIB037 by intravenous infusion.
  Interventions: Drug: BIIB037
- Placebo (Placebo Comparator): A single dose of placebo matching BIIB037 by intravenous infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BIIB037 — Participants receive a single dose of BIIB037 by intravenous (IV) infusion in cohorts assigned to the following ascending doses: .03 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg, and 60 mg/kg.
  Other Names: Aducanumab; fully human IgG1 anti-Aβ mAb
  Arms: BIIB037
Other: Placebo — Participants receive a single dose of matching BIIB037 placebo by intravenous (IV) infusion.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of a range of BIIB037 doses administered as single intravenous (IV) infusions in participants with mild to moderate Alzheimer's Disease (AD). Secondary objectives of this study in this study population are to assess the pharmacokinetics(PK) and to evaluate the immunogenicity of BIIB037 after single-dose administration.

DETAILED DESCRIPTION:
BIIB037 is an investigational product being developed as a treatment for Alzheimer's disease (AD). BIIB037 is a fully human immunoglobulin gamma 1 (IgG1) monoclonal antibody that is selective for the fibrillar form of beta amyloid (Aß).

ELIGIBILITY:
Key Inclusion Criteria:

* Must be ambulatory
* Must have a clinical diagnosis of Alzheimer's Disease (AD) consistent with the following:

  1. Probable Alzheimer's Disease (AD), according to National Institute of Neurological and Communicative Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria [McKhann et al. 1984].
  2. Dementia of Alzheimer's type, according to Diagnostic and Statistical Manual of Mental Disorders-Text Revision (DSM IV TR) criteria [American Psychiatric Association 2000]
* Subject (or subject's permanent caregiver) has the ability to understand the purpose and risks of the study and provide signed and dated informed consent (or assent) and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Must have a Mini Mental State Examination (MMSE) score of 14 to 26 inclusive.

Key Exclusion Criteria:

* Any medical or neurological condition other than Alzheimer's Disease (AD) that in the opinion of the Investigator could be a contributing cause of the subject's dementia (e.g., medication use, vitamin B12 deficiency, abnormal thyroid function, stroke or other cerebrovascular condition, diffuse Lewy body disease, head trauma).
* History within the past 6 months or evidence of clinically significant psychiatric illness (e.g., major depression, schizophrenia, or bipolar affective disorder).
* Subject currently lives in a nursing home.
* Blood donation (1 unit or more) within the 1 month prior to Screening
* Participation in any other drug, biologic, device, or clinical study or treatment with any investigational drug or approved therapy for investigational use within 30 days (or 5 half lives, whichever is longer) prior to Screening, and/or participation in any other clinical study involving experimental medications for AD within the 60 days (or 5 half lives, whichever is longer) prior to Screening.
* Any contraindications to having a brain Magnetic Resonance Imaging (MRI) e.g., pacemaker; Non-Magnetic Resonance Imaging (MRI)-compatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months
  Incidence and nature of adverse events (AEs) and serious adverse events (SAEs). Significant assessments reported as AEs or SAEs include clinical laboratory assessments and vital signs, physical and neurological examination, 12-lead electrocardiogram (ECG), and brain MRI findings (including the occurrence of vasogenic edema and incident hemorrhage).

SECONDARY OUTCOMES:
Area Under the Curve from Time Zero Extrapolated to Infinity [AUC0-∞] | 6 months
Area Under the Curve from Time 0 to Time of the Last Measurable Concentration [AUC0-tlast] | 6 months
Maximum Concentration [Cmax] of BIIB037 | 6 Months
Time to Cmax [Tmax] | 6 Months
Elimination Half-life [t1/2] | 6 Months
Clearance [Cl] | 6 Months
Incidence of Anti-BIIB037 Antibodies in Serum | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - Brain Matters Research, Delray Beach, Florida
  - Compass Research, LLC, Orlando, Florida
  - Insight Clinical Trials, LLC, Beachwood, Ohio

REFERENCES:
- [Derived] Ferrero J, Williams L, Stella H, Leitermann K, Mikulskis A, O'Gorman J, Sevigny J. First-in-human, double-blind, placebo-controlled, single-dose escalation study of aducanumab (BIIB037) in mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2016 Jun 20;2(3):169-176. doi: 10.1016/j.trci.2016.06.002. eCollection 2016 Sep. PMID 29067304